CLINICAL TRIAL: NCT07235709
Title: Effect of Agalsidase Alfa on Cardiac Inflammation in Patients With Fabry Disease: A [18F]-FDG PET-CMR Study (ESCAPE-FABRY Trial)
Brief Title: Effect of Agalsidase Alfa on Cardiac Inflammation in Patients With Fabry Disease: A [18F]-FDG PET-CMR Study
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2025-1005
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fabry's disease: atients aged 15-75 years with Fabry disease confirmed by enzyme assay and gene test

SUMMARY:
This is a prospective observational study. All patients will initiate and maintain treatment with agalsidase alfa during the study period. All patients will receive a full standard of care concomitant medication for the treatment of their cardiac condition. Twenty-five patients with genetically confirmed Anderson-Fabry disease will undergo PET-CMR at baseline and after 12 months of treatment with Agalsidase Alfa for follow-up.

DETAILED DESCRIPTION:
Visit 1. Screening At screening, for potential eligible patients, after obtaining their informed consent, inclusion/exclusion criteria will be reviewed and enrollment will be determined. Demography (date of birth, gender), prior and concomitant medication and relevant medical history will be recorded. Height, body weight, vital signs, and laboratory assessments will be needed. Women of childbearing potential will be tested for pregnancy.

Visit 2. Baseline Study At visit 2, subjects have following baseline evaluations performed

* Laboratory test: CBC+PLT, WBC Differential Count, Routine Chemistry (Calcium, Inorganic P, BUN, Creatinine, Fasting Glucose, Cholesterol, Total Protein, Albumin, Total. Bilirubin, Alkaline Phosphatase, AST, ALT), Electrolyte(Na, K, Cl), Lipid profile(Triglyceride, HDL-Cholesterol, LDL-Cholesterol), Plasma Lyso-GB3, NT-proBNP, Troponin T, high-sensitive C-reactive protein, ESR, Interleukin 6, Soluble urokinase plasminogen activator receptor (suPAR), monocyte chemoattractant protein-1(MCP-1), matrix metalloprotease-9(MMP-9), Tumor necrosis factor receptor 2(TNFR2), Urinalysis with Microscopy, Urine test(Microalbumin, Creatinine, Microprotein,Total), Anti-body testing for agalsidase alfa
* Concomitant medication
* Vital signs, weight
* 12-lead ECG
* QOL questionnaire
* PET-CMR
* MIBG cardiac scintigraphy (not mandatory)
* Conventional Echocardiography including strain imaging

Two-dimensional echocardiography Standard 2-dimensional measurements (LV diastolic and systolic dimensions, ventricular septum and posterior wall thickness, left atrial volume, and LV outflow tract diameter) will be obtained with the patients in the left lateral position. LV ejection fraction (EF) will be calculated by the Simpson's method. From the apical window, a 1- to 2-mm pulsed Doppler sample volume will be placed at the mitral valve tip and mitral flow velocities from 5-10 cardiac cycles will be recorded. Mitral inflow velocities are traced and the following variables will be obtained: peak velocity of early (E) and late (A) filling, and deceleration time of E-wave velocity. Stroke volume (SV) will be measured from LV outflow tract diameter and pulse-wave Doppler signal as previously described. Mitral annular velocity will be measured by Doppler tissue imaging using pulse-wave Doppler mode. The filter will be set to exclude high frequency signal, and the Nyquist limit will be adjusted to a range of 15-20 cm/s. Gain and sample volume will be minimized to allow for a clear tissue signal with minimal background noise. Early diastolic (E') and systolic (S') velocities of the mitral annulus will be measured from the apical 4-chamber view with a 2- to 5-mm sample volume placed at the septal corner of the mitral annulus. All data will be stored digitally and measurements will be taken at the completion of each study. Two-dimensional echocardiographic images from apical views at rest will be acquired, digitized, recorded, and analyzed for the wall motion analysis. Using a dedicated software package (EchoPAC PC), LV-GLS, LV global circumferential strain (LV-GCS), and LV global radial strain (LV-GRS) will be calculated automatically. 2D strain is a non-Doppler-based method for the evaluation of systolic strain using standard 2D acquisitions. LV-GLS strain will be assessed in three apical views, and LV-GCS and LV-GRS will be assessed in three levels of parasternal short-axis views. Left atrial (LA) strain also will be assessed by the same software.

Positron Emission Tomography - Cardiac Magnetic Resonance Imaging (PET-CMR) The PET-CMR procedure will be conducted prior to and within 12 months after initiating Enzyme Replacement Therapy (ERT). All patients are instructed to take a high-fat low-carbohydrate diet the day prior with overnight fast. Administer intravenous unfractionated heparin at a dose of 50 units/kg approximately 15 minutes before the intravenous injection of 10-12 mCi of 18F-FDG. This method is suitable for patients without any bleeding tendencies. After a 90-minute uptake period, cardiac and partial whole body PET images (cerebellum to mid-thigh) are acquired.The F-18 FDG study commences following an oral glucose load of 50 grams, administered one hour prior to injecting 370 MBq of F-18 FDG. A simultaneous cardiac PET/MR study is conducted on an integrated PET/MR scanner (Biograph mMR, Siemens Healthcare, Erlangen, Germany) beginning one hour after the tracer injection. Initially, a standard Dixon sequence is acquired for attenuation correction. Subsequently, comprehensive cardiac MR (CMR) sequences are performed. These include steady-state free precession cine imaging in two-chamber, three-chamber, and four-chamber views, as well as in short-axis images, to ensure detailed cardiac assessment. MR perfusion imaging is performed following gadolinium contrast infusion, and post-contrast late gadolinium enhancement (LGE) studies are executed for detailed tissue characterization. Static F-18 FDG myocardial PET imaging is acquired concurrently during the MRI scans, utilizing list mode for a duration of 30 minutes. The maximal myocardial thickness is noted as 30 mm at end-diastole on cine MRI. The first-pass MR perfusion imaging indicates reduced myocardial blood flow, while patchy F-18 FDG defect areas correspond to regions of LGE, indicative of myocardial fibrosis. Correlate findings from PET and CMR to gain for evaluation of Fabry cardiomyopathy, including assessment of myocardial viability, detection of ischemia, and characterization of tissue.

123I-meta-iodobenzylguanidine scintigraphy The 123I-meta-iodobenzylguanidine (MIBG) scintigraphy will be conducted prior to and within 12 months after initiating ERT. MIBG scintigraphy is expected to provide information to determine whether cardiac sympathetic nerve dysfunction is present in patients with Fabry disease. (8, 9) Because it is reported that decreased MIBG uptake in the inferolateral wall compared with the anteroseptum in patients with LGE of the inferolateral wall in patients with Fabry cardiomyopathy. Moreover, MIBG imaging may play a unique role in assessing the risk of developing ventricular arrhythmia and sudden cardiac death (SCD).

MIBG cardiac imaging will be conducted in according to the current standard.(10, 11) An intravenous dose of 222 MBq 123I-MIBG will be administered by slow (1-2 min) injection through a peripheral venous cannula after thyroid protection via oral intake of 300 mg of potassium perchlorate. All images will be acquired using a Optima NM/CT 640 gamma camera (GE Healthcare, Milwaukee, WI, USA) at 15 (early) and 180 minutes (late) post injection of MIBG. Planar images will be acquired with a low energy high-resolution sensitivity (LEHRS) collimator, 159 keV ± 10% energy window, 256 × 256 image matrix, and zoom of 1.0 (pixel size 2.21 mm) for 1.5 minutes. SPECT images will be acquired over a 180° orbit from the right anterior oblique to left posterior oblique positions with LEHRS collimators, 159 keV ± 10% energy window, 64 × 64 image matrix, zoom of 1.28 (pixel size 6.9 mm) and 60 projections at 17 seconds per projection. The heart-to-mediastinum (H/M) ratio of MIBG uptake and the MIBG defect size will be assessed. MIBG scintigraphy will be conducted for a secondary endpoint and is not mandatory for all patients. It is only performed on patients who have provided consent for the test.

Visit 3. Treatment week 12 At visit 3, subjects have following evaluations performed

* Concomitant medication
* Laboratory test: CBC+PLT, WBC Differential Count, Routine Chemistry (Calcium, Inorganic P, BUN, Creatinine, Fasting Glucose, Cholesterol, Total Protein, Albumin, Total. Bilirubin, Alkaline Phosphatase, AST, ALT), Electrolyte(Na, K, Cl), Plasma Lyso-GB3, Urinalysis with Microscopy
* Vital signs, weight
* 12-lead ECG
* QOL questionnaire
* Adverse events monitoring Visit 4. Treatment week 24 At visit 4, subjects have following evaluations performed
* Concomitant medication
* Laboratory test: CBC+PLT, WBC Differential Count, Routine Chemistry (Calcium, Inorganic P, BUN, Creatinine, Fasting Glucose, Cholesterol, Total Protein, Albumin, Total. Bilirubin, Alkaline Phosphatase, AST, ALT), Electrolyte(Na, K, Cl), Plasma Lyso-GB3, NT-proBNP, Troponin T, ESR, Urinalysis with Microscopy
* Vital signs, weight
* 12-lead ECG
* QOL questionnaire
* Adverse events monitoring

Visit 5. Treatment week 52 (End of study) At visit 5, subjects have following final evaluations performed

* Laboratory test: CBC+PLT, WBC Differential Count, Routine Chemistry (Calcium, Inorganic P, BUN, Creatinine, Fasting Glucose, Cholesterol, Total Protein, Albumin, Total. Bilirubin, Alkaline Phosphatase, AST, ALT), Electrolyte(Na, K, Cl), Lipid profile(Triglyceride, HDL-Cholesterol, LDL-Cholesterol), Plasma Lyso-GB3, NT-proBNP, Troponin T, high-sensitive C-reactive protein, ESR, Interleukin 6, Soluble urokinase plasminogen activator receptor (suPAR), monocyte chemoattractant protein-1(MCP-1), matrix metalloprotease-9(MMP-9), Tumor necrosis factor receptor 2(TNFR2), Urinalysis with Microscopy, Urine test(Microalbumin, Creatinine, Microprotein,Total), Anti-body testing for agalsidase alfa
* Concomitant medication
* Vital signs, weight
* 12-lead ECG
* QOL questionnaire
* PET-CMR
* MIBG cardiac scintigraphy (not mandatory)
* Conventional Echocardiography including strain imaging
* Adverse events monitoring

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15-75 years with Fabry disease confirmed by enzyme assay and gene test
* Patients have not undergone ERT for more than 12 months or patients have not used Agalsidase Alfa in the last 12 months.
* Patients who have cardiac involvement of Fabry disease (end diastolic maximal wall thickness ≥ 12mm on echocardiography or CMR, decreased native T1 value on CMR, unexplained distinct diastolic dysfunction, unexplained decreased global longitudinal strain on 2D strain echocardiography, or biopsy-proven cardiac involvement)
* Patients provided written informed consent to participate in this study
* The patient, or patient's legally authorized representative(s), if applicable, understands the nature, scope, and possible consequences of the study and has provided written informed consent that has been approved by the Institutional Review Board/Independent Ethics Committee
* The patient must be sufficiently cooperative to participate in this clinical study as judged by the investigator.

Exclusion Criteria:

* Contraindication for enzyme replacement treatment with Agalsidase Alfa
* Patients have previously been treated with Agalsidase Alfa for > 12 months
* Patients unable to undergo PET-CMR due to any condition
* Patients who are pregnant
* Patients who have active malignancy
* Subject who the investigator deems inappropriate to participate in this study

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 15 ~ 75 years with Fabry disease confirmed by enzyme assay and gene test
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of ERT with Agalsidase Alfa on change of myocardial inflammation in patients with Fabry's cardiomyopathy using PET-CMR. | 1 year
  To evaluate the impact of ERT with Agalsidase Alfa on change of myocardial inflammation in patients with Fabry's cardiomyopathy using PET-CMR.

SECONDARY OUTCOMES:
To evaluate myocardial inflammation in patients with Fabry disease before ERT | 1 year
  To evaluate myocardial inflammation in patients with Fabry disease before ERT
To evaluate myocardial inflammation in patients with Fabry disease during ERT | 1 year
  To evaluate myocardial inflammation in patients with Fabry disease during ERT
To evaluate myocardial fibrosis in patients with Fabry disease before ERT | 1 year
  To evaluate myocardial fibrosis in patients with Fabry disease before ERT
To evaluate myocardial fibrosis in patients with Fabry disease during ERT | 1 year
  To evaluate myocardial fibrosis in patients with Fabry disease during ERT
To evaluate cardiac cardiac sympathetic nerve dysfunction during ERT | 1 year
  To evaluate cardiac cardiac sympathetic nerve dysfunction during ERT

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided